CLINICAL TRIAL: NCT01430910
Title: A Phase I, 2-Part, Open-Label, Pharmacokinetic and Drug-Drug Interaction Study of CAZ104 (Avibactam and Ceftazidime in Healthy Subjects)
Brief Title: A Study to Assess the Levels of Two Antibiotics in the Blood When Given Together and Separately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00011
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Phase 1; open label; ceftazidime; pharmacokinetics; urinary tract infection; intra-abdominal infection
MeSH Terms: conditions — Urinary Tract Infections; Intraabdominal Infections | interventions — avibactam; Ceftazidime

ARMS (3):
- 1 (Experimental): CAZ104 (2000mg Ceftazidime/500mg Avibactam)
  Interventions: Drug: CAZ104
- 2 (Active Comparator): 500mg Avibactam
  Interventions: Drug: Avibactam
- 3 (Active Comparator): 2000mg Ceftazidime
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: CAZ104 — IV infusion
  Arms: 1
Drug: Avibactam — IV infusion
  Arms: 2
Drug: Ceftazidime — IV infusion
  Arms: 3

SUMMARY:
This is a randomised study divided into 2 parts. Part A investigates the effect of prolonged dosing (ten days) with Avibactam and Ceftazidime when given together and how this will effect how much Avibactam and Ceftazidime enters the blood. Part B investigates how much Avibactam (NXL104) and Ceftazidime enter the blood when Avibactam and Ceftazidine are given separately or together intravenously.

DETAILED DESCRIPTION:
A Phase I, 2-Part, Open-Label, Pharmacokinetic and Drug-Drug Interaction Study of CAZ104 (Avibactam and Ceftazidime in Healthy Subjects)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male and female subjects aged 18 to 50 years with veins suitable for cannulation or repeated venepuncture; female subjects must be postmenopausal or surgically sterile. Female subjects must have a negative pregnancy test at screening and on admi
* Male subjects should be willing to use barrier contraception ie, condoms, from dosing to 3 months after dosing with the IP (investigational product).
* Have a body mass index (BMI) between 19 and 30 kg/m2
* As judged by the Investigator, all the subjects must be able to understand and be willing to comply with study procedures, restrictions and requirements

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to avibactam, ceftazidime, and/or excipients
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP Prolonged QTcF (>450 ms) or shortened QTcF (<350 ms) or a family history of long QT syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including maximum plasma concentration (Cmax) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including time of Cmax (tmax) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including minimum plasma concentration (Cmin) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including time of Cmin (tmin) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including last quantifiable plasma concentration (Clast) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including time of Clast (tlast) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including average plasma concentration during a dosing interval (Cavg) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including fluctuation index | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including area under the curve of plasma drug concentration (AUC) - time curve from zero to the time of the last quantifiable concentration | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including AUC, Day 1 only | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including AUC during the dosing interval [AUC(0-τ)] | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including terminal half-life (t1/2) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including systemic plasma clearance (CL) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including volume of distribution at steady state (Vss) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including volume of distribution at the terminal phase (Vz) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including accumulation ratio for Cmax and AUC(0-τ) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Plasma pharmacokinetic variables will be measured including linearity index | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Urine pharmacokinetic variables will be measured including amount of drug excreted unchanged into urine from zero to time t [Ae(0-t)] | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Urine pharmacokinetic variables will be measured including fraction of dose excreted unchanged into urine (fe; % dose) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Avibactam. Urine pharmacokinetic variables will be measured including renal clearance (CLR) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Cmax | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including tmax | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Cmin | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including tmin | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Clast | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including tlast | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Cavg | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including fluctuation index | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including AUC(0-t) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including AUC, Day 1 only | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including AUC(0-τ) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including t1/2 | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including CL | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Vss | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including Vz | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including accumulation ratio for Cmax and AUC(0-τ) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Plasma pharmacokinetic variables will be measured including linearity index | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Urine pharmacokinetic variables will be measured including Ae(0-t) | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Urine pharmacokinetic variables will be measured including fe; % dose | Up to 24 hours post last dose
Part A: Single- and multiple-dose pharmacokinetics of Ceftazidime. Urine pharmacokinetic variables will be measured including CLR | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Cmax | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including tmax | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Cmin | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including tmin | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Clast | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including tlast | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Cavg | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including fluctuation index | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including AUC(0-t) | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including AUC, Day 1 only | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including AUC(0-τ) | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including t1/2 | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including CL | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Vss | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including Vz | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including accumulation ratio for Cmax and AUC(0-τ) | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Plasma pharmacokinetic variables will be measured including linearity index | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Urine pharmacokinetic variables will be measured including Ae(0-t) | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Urine pharmacokinetic variables will be measured including fe; % dose | Up to 24 hours post last dose
Part B: Pharmacokinetics of co-administering Avibactam plus Ceftazidime (CAZ104) compared to administration of the individual components. Urine pharmacokinetic variables will be measured including CLR | Up to 24 hours post last dose

SECONDARY OUTCOMES:
To assess safety and tolerability of Avibactam by assessment of Adverse events | Up to 24 hours post last dose
To assess safety and tolerability of Avibactam by clinical laboratory assessments | Up to 24 hours post last dose
To assess safety and tolerability of Avibactam by assessment of vital signs | Up to 24 hours post last dose
To assess safety and tolerability of Avibactam by assessment of safety electrocardiogram | Up to 24 hours post last dose
To assess safety and tolerability of Avibactam by assessment of physical examination | Up to 24 hours post last dose
To assess safety and tolerability of Avibactam by assessment of withdrawn | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by assessment of Adverse events | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by clinical laboratory assessments | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by assessment of vital signs | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by assessment of safety electrocardiogram | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by assessment of physical examination | Up to 24 hours post last dose
To assess safety and tolerability of Ceftazidime by assessment of withdrawn | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by assessment of Adverse events | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by clinical laboratory assessments | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by assessment of vital signs | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by assessment of safety electrocardiogram | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by assessment of physical examination | Up to 24 hours post last dose
To assess safety and tolerability of CAZ104 by assessment of withdrawn | Up to 24 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Mirjana Kujacic, MD, Study Chair — AstraZeneca Research and DevelopmentSE-431 83 Mölndal Sweden; Leonard Siew, MBCHB, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital 6 Newcomen St London SE1 1YR United Kingdom; Paul Newell, MD, Study Director — AstraZeneca R&D Alderly Park, Mereside SK 104 TG Macclesfield, Cheshire United Kingdom
Locations (1):
- Research site, London, United Kingdom

REFERENCES:
- [Background] Das S, Li J, Armstrong J, Learoyd M, Edeki T. Randomized pharmacokinetic and drug-drug interaction studies of ceftazidime, avibactam, and metronidazole in healthy subjects. Pharmacol Res Perspect. 2015 Oct;3(5):e00172. doi: 10.1002/prp2.172. Epub 2015 Aug 25. PMID 26516584
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- See also: Redaction of D4280C00011 Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1457&filename=Redaction%20of%20D4280C00011%20Protocol.pdf